CLINICAL TRIAL: NCT04811768
Title: Comparative Clinical and Histological Investigation of Graft Integration Following Piezosurgically Retrieved Lateral Bony Wall Repositioning in Maxillary Sinus Floor Augmentation - Prospective Randomized Controlled Study
Brief Title: Lateral Bony Wall Repositioning in Maxillary Sinus Floor Augmentation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: NSK Europe GmbH (Industry); Botiss Medical AG (Other); Institut Straumann AG (Industry); Dicomlab Kft. (Unknown); Hungarian Human Resources Development Operational Program (EFOP-3.6.2-16-2017-00006) (Unknown); Excellence Program of the Ministry for Innovation and Technology in Hungary (Unknown)
Responsible Party: Principal Investigator, Balint Molnar, Dr. Balint Molnar DMD, PhD, associate professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sinus-Semmelweis-Perio
Record Dates: First submitted 2021-03-09; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Maxillary Sinus Augmentation
Keywords: maxillary sinus; xenogeneic graft; collagen membrane; lateral bony wall repositioning; piezoelectric surgery
MeSH Terms: interventions — Sinus Floor Augmentation

STUDY DESIGN:
Intervention Model Description: 40 patients underwent sinus floor augmentation - 20 patients treated by bony wall repositioning, 20 patients treated by collagen membrane coverage
Who Masked: Outcomes Assessor
Masking Description: Histology analysis was performed blinded, randomization sequence was revealed after histomorphometry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bony wall group (Experimental): In the bony wall group, following piezosurgery the retrieved bony wall was repositioned.
  Interventions: Procedure: Maxillary sinus augmentation
- Collagen membrane group (Experimental): In the collagen membrane group, the lateral window was created by rotary instruments, covered via a native collagen membrane (collprotect, botiss biomaterials GmbH, Zossen, Germany).
  Interventions: Procedure: Maxillary sinus augmentation

INTERVENTIONS:
Procedure: Maxillary sinus augmentation — The surgery was performed under local anaesthesia in both groups, lateral window preparation and window coverage was carried out based on randomization.
  Other Names: Sinus lift

SUMMARY:
The aim of the present prospective randomized controlled study is to clinically and histologically investigate the safety and efficacy of bony wall repositioning compared to rotary window preparation with membrane coverage in maxillary sinus floor augmentation.

DETAILED DESCRIPTION:
40 patients were randomly divided in two study groups after radiological and clinical evaluation. Both groups received bone grafting by a xenogeneic bone substitute (BSM, cerabone, botiss biomaterials GmbH, Zossen, Germany) using the lateral approach. In the bony wall group (BW), following piezosurgery the retrieved bony wall was repositioned. In the collagen membrane group (CM), the lateral window was created by rotary instruments, covered via a native collagen membrane (collprotect, botiss biomaterials GmbH, Zossen, Germany). After 6 months, biopsies were taken to analyze both approaches in terms of new bone formation. Duration of treatment, the number of perforations, postoperative patient discomfort were registered. Established histopathological analysis and histomorphometrical measurements to analyze the tissue reactions and the tissue distribution, i.e., the fractions of newly formed bone tissue (NB), of remaining bone substitute material (BSM) and connective tissue (CT), were conducted.

ELIGIBILITY:
Inclusion Criteria:

* at least one missing maxillary premolar or molar
* at least 7 mm crestal bone width confirmed by preoperative ConeBeam Tomography (CBCT)
* maximally 5 mm residual bone height at the sinus floor confirmed by preoperative ConeBeam Tomography (CBCT)
* full mouth plaque and bleeding scores (FMPS and FMBS) <20%
* satisfactory patient compliance (e.g. to participate in follow-up procedures)
* signed informed consent.

Exclusion Criteria:

* clinically relevant diseases (e.g.: diabetes, rheumatism cancer)
* untreated periodontitis
* systemic steroid use
* bisphosphonate use
* acute or chronic inflammatory processes
* previous endoscopic sinus surgery
* previous sinus floor elevation
* GBR-treatment at the study site
* GTR-treatment at the study site
* tooth removal within 6 weeks prior to surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Duration of surgery | During smaxillary sinus augmentation
  Recorded in minutes

SECONDARY OUTCOMES:
Duration of lateral window preparation | During maxillary sinus augmentation
  Recorded in minutes
Duration of mucosa preparation | During maxillary sinus augmentation
  Recorded in minutes
Visual Analog Scale (Minimum value 0, Maximum value 100, the higher the worse) | 12 hours postoperatively
  Measurement of patient discomfort
Visual Analog Scale (Minimum value 0, Maximum value 100, the higher the worse) | 1 day postoperatively
  Measurement of patient discomfort
Postoperative Edema Score | 2 days postoperatively
  Measurement of swelling
Postoperative Edema Score | 3 days postoperatively
  Measurement of swelling
Histomorphometrical analysis | Following reentry 6 months after maxillary sinus augmentation
  Percentage of newly formed bone, bone substitute and connective tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Department of Periodontology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molnar B, Jung AK, Papp Z, Martin A, Orban K, Prohl A, Jung O, Barbeck M, Windisch P. Comparative analysis of lateral maxillary sinus augmentation with a xenogeneic bone substitute material in combination with piezosurgical preparation and bony wall repositioning or rotary instrumentation and membrane coverage: a prospective randomized clinical and histological study. Clin Oral Investig. 2022 Aug;26(8):5261-5272. doi: 10.1007/s00784-022-04494-x. Epub 2022 May 20. PMID 35593928